CLINICAL TRIAL: NCT01001468
Title: A Randomized, Double-Blind, 12-Week, Dose-Ranging Placebo-Controlled Study to Evaluate the Efficacy and Safety of Oral VB-201 in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Study to Assess VB-201 in Patients With Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vascular Biogenics Ltd. operating as VBL Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VB-201-006
Record Dates: First submitted 2009-10-20; First posted 2009-10-26 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Active Plaque Psoriasis
Keywords: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — 1-palmityl-2-(4-carboxybutyl)-sn-glycero-3-phosphocholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VB-201 20 mg (Experimental)
  Interventions: Drug: VB-201
- VB-201 80 mg (Experimental)
  Interventions: Drug: VB-201
- Placebo (Placebo Comparator): Single daily dose of oral placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: VB-201 — Single daily dose of oral VB-201 20 mg
  Arms: VB-201 20 mg
Drug: VB-201 — Single daily dose or oral VB-201 80 mg
  Arms: VB-201 80 mg
Other: Placebo — Single daily dose of oral placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy, safety and tolerability of VB-201 as compared with placebo on measures of disease activity in patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Patients, ≥18 to ≤75 years of age, who have a diagnosis of chronic plaque psoriasis for at least 6 months
* Non-anorexic subjects with a BMI ≥20
* Psoriasis Area and Severity Index (PASI) score of ≥12
* Plaque psoriasis covering ≥10% of body surface area (BSA)
* Psoriasis severity at least moderate, scoring at least 3 on the 0 to 5 point Physician Global Assessment (PGA) scale

Exclusion Criteria:

* The subject presents with the predominant type of psoriasis as guttate, erythrodermic, inverse, pustular or palmo-plantar or an unstable form of psoriasis
* The subject has not undergone wash-out periods of sufficient duration for the following treatments at Baseline: Topical psoriasis treatments; Systemic, oral or injected, psoriasis treatments; Phototherapy
* The subject anticipates getting enough ultra-violet light during the study to cause psoriasis to improve
* The subject has a known allergy or sensitivity to the study treatment(s) or to any of the excipients contained in the study drug formulation
* History of cancer, the exception is skin cancer
* Has a clinically significant systemic infection within 30 days of Day 0, or a history or presence of recurrent or chronic infection
* Evidence of tuberculosis as indicated by a positive tuberculin skin test or a quantiferon test in subjects known to have a + PPD and a negative chest x-ray at screening
* History of clinically significant hypoglycemia
* Subjects with currently active peptic ulcer / gastroesophageal reflux disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2009-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Improvement in the Psoriasis Area and Severity Index(PASI 75)from baseline at Week 12 | 20 weeks

SECONDARY OUTCOMES:
Change in PGA (Physician Global Assessment) scores from baseline to Week 12 | 20 weeks
Change in Patient Psoriasis Global Assessment scores from baseline to Week 12 | 20 weeks
Change in affected Body Surface Area (BSA) from baseline to Week 12 | 20 weeks
Measurement of improvement in the PASI (50) from baseline at Week 12 | 20 weeks

CONTACTS AND LOCATIONS:
Locations (18):
- United States (10):
  - Alexa Kimball, MD, Massachusetts General and Brigham and Women's Hospital, Boston, Massachusetts
  - Mark Amster, MD, Boston Clinical Trials, Boston, Massachusetts
  - David Greenstein, MD, ActivMed Practices and Research, Haverhill (Boston), Massachusetts
  - Craig Leonardi, MD, Central Dermatology, St Louis, Missouri
  - Bruce Strober, MD, New York University Medical Center, Dermatologic Associates, New York, New York
  - Gary Goldenberg, MD, Mount Sinai School of Medicine, New York, New York
  - Julian MacKay Wiggan, MD, Columbia University Medical Center, New York, New York
  - Steven Cohen, MD, Montefiore Medical Center, Dermatology, New York, New York
  - Joseph D. Sutton, MD, PC, Suffern, New York
  - Kristina Callis-Duffin, MD, University of Utah, Salt Lake City, Utah
- Germany (7):
  - Sandra Philipp, MD, Charité Campus Mitte, Universitaetsmedizin Berlin, Berlin
  - Rolf Dominicus, MD, Praxisklinik und Gemeinschaftspraxis, Dülmen
  - Bernhard Homey, MD, Universitaetsklinikum Duesseldorf, Düsseldorf
  - Diamant Thaci, MD, Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt
  - Ulrich Mrowietz, MD, Universitaetsklinikum Schleswig-Holstein, Kiel
  - Michael Sebastian, MD, SCIDerm GmbH, Mahlow
  - Rudolf Schopf, MD, Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz KoeR, Mainz
- Professor Michael David, MD, Beilinson Hospital, Petach Tikvah, Israel